CLINICAL TRIAL: NCT00702221
Title: A Randomised, Double Blind, Placebo Controlled Study of the Efficacy and Safety of Angiotensin Therapeutic Vaccine (ATV) in Subjects With Mild to Moderate Hypertension
Brief Title: Safety and Efficacy Study of Angiotensin Therapeutic Vaccine in Subjects With Mild to Moderate Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Dose limiting adverse effects
Sponsor: BTG International Inc. (Other)
Collaborators: Encorium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR002-CLN-pro008
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-04

CONDITIONS: Hypertension; Cardiovascular Disease
Keywords: high blood pressure; vaccines
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATV with CoVaccine HT™ (Experimental): Angiotensin Therapeutic Vaccine with CoVaccine HT™ adjuvant (an ingredient that may improve the immune response of the vaccine)
  Interventions: Biological: Angiotensin Therapeutic Vaccine plus CoVaccine HT™ adjuvant
- CoVaccine HT™ adjuvant alone (Placebo Comparator): CoVaccine HT™ adjuvant alone
  Interventions: Biological: CoVaccine HT™ adjuvant

INTERVENTIONS:
Biological: Angiotensin Therapeutic Vaccine plus CoVaccine HT™ adjuvant — Angiotensin Therapeutic Vaccine plus CoVaccine HT™ adjuvant given as 3 separate intramuscular injections into the arm, 21 days apart
  Arms: ATV with CoVaccine HT™
Biological: CoVaccine HT™ adjuvant — Given as three separate intramuscular injections into the arm, 21 days apart
  Arms: CoVaccine HT™ adjuvant alone

SUMMARY:
Angiotensin Therapeutic Vaccine (ATV), which contains the novel adjuvant, CoVaccine HT™ , is being developed for the treatment of high blood pressure (hypertension), a major risk factor for serious diseases such as heart attacks and strokes. Many patients with high blood pressure fail to take their medicines as prescribed because they generally feel well, which often results in poor control of the condition. As a result, it is estimated that about 70% patients with hypertension do not have their blood pressure adequately controlled despite advances in the treatment of high blood pressure.

The main aim of this study is to find out if an injection of ATV given in the arm once every 3 weeks on 3 occasions results in lowering overall blood pressure measurements throughout the day. The other aims are to find out if ATV is safe and to see how well it is tolerated

DETAILED DESCRIPTION:
One of the causes of hypertension is overactivity of the renin angiotensin system, the main mechanism by which the human body regulates its sodium and water balance. An enzyme called renin cleaves a peptide from the protein angiotensinogen, releasing angiotensin I (AI), which is then converted to a peptide hormone called angiotensin II (AII) by the angiotensin converting enzyme (ACE). Angiotensin II is a hormone which is a powerful vasoconstrictor and increases blood flow to vital organs. Angiotensin Therapeutic Vaccine acts by inducing antibodies which bind to angiotensin, so suppressing its actions.

ATV may offer a way of improving control of blood pressure by increasing patient compliance with treatment. Infrequent vaccinations may provide a sustained reduction in blood pressure and afford a desirable, slow onset of action. Such a vaccine could provide an adjunct to and possibly a replacement for existing therapy in some patients, particularly where patient compliance is likely to be a problem.

This study will determine if three injections of ATV given over the period of six weeks will reduce daytime BP as measured by ambulatory blood pressure monitoring.

The study is split into 2 stages Stage A and Stage B.

The rationale behind Stage A is to closely evaluate the safety and tolerability of ATV in a small number of subjects prior to enroling the majority of subjects into the remaining portion of the study. Stage A will include a minimum of 12 subjects who will receive each of their three injections at a dedicated Phase 1 facility with access to critical care facilities.

Based on the safety profile of the stage A subjects, a recommendation will be made by an independent Data Safety Monitoring Committee on whether to proceed to Stage B.

Stage B will include approximately 112 subjects. As safety and tolerability will have been closely assessed in Stage A, Stage B subjects will be monitored less closely and will be recruited from a number of sites in the UK.

ELIGIBILITY:
Inclusion Criteria (at randomisation):

1. Competent to provide written informed consent
2. 35-70 years old
3. Body Mass Index (BMI) 19 to 33 kg/m2
4. Mild to moderate hypertension per British Hypertension Society (BHS) Guidelines BHS-IV based on the following criteria of sitting blood pressure for subjects without diabetes or renal dysfunction.
5. Average sitting morning DBP 90 to 109 mmHg and SBP 140 to 179 mmHg and have responded positively to a quinapril challenge.

Principal exclusion criteria:

1. Women of childbearing potential: defined to be not surgically sterile and <2 y post-menopausal
2. Average sitting SBP of >180 mmHg or DBP of >110 mmHg.
3. A BP difference between left and right arm greater than 20 mmHg for SBP and 10 mmHg for DBP which is present on 3 consecutive readings.
4. Left ventricular (LV) systolic dysfunction as evidenced by a known LV ejection fraction <40% or symptomatic congestive heart failure requiring treatment.
5. HbA1c >7.0% or a history of Type 1 or Type 2 diabetes.
6. Haemoglobin <12 g/dL at Screening.
7. Hypo- or hyperthyroidism
8. Serum alanine aminotransferase or aspartate aminotransferase >2X ULN.
9. Other identifiable secondary causes of hypertension
10. Myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 6 months of Screening.
11. Bradycardia <50 beats per minute at rest in the supine position prior to randomisation.
12. Have sick sinus syndrome or second or third degree atrioventricular block, chronic atrial fibrillation or recurrent atrial tachyarrhythmia (including paroxysmal atrial tachycardia), history of recurrent ventricular tachycardia, or symptomatic bradycardia.
13. Implanted pacemakers or cardioverter defibrillator.
14. Haemodynamically significant valvular heart disease.
15. History of renal dysfunction and/or estimated glomerular filtration rate <60 mL/min/1.73 m2.
16. Diagnosis or recurrence of malignancy within the past 3 years, with the exception of basal cell carcinoma of the skin or in situ carcinoma of the cervix.
17. Sleep apnea unless a recent (within 30 days of Screening) sleep study demonstrates no recordings of arterial oxygen saturation (SaO2) <90%, treated or untreated, at any time during the Screening Period.
18. Perform alternating shift or night work.
19. Not on stable doses of all concomitant medications for a minimum of 4 weeks prior to Screening, and subjects treated with any of the following prohibited medications:

    * Oral corticosteroids within 3 months of Screening.
    * Acetylsalicylic acid in excess of 325 mg per day.
    * Chronic stable or unstable use of non-steroidal anti-inflammatory drugs (NSAIDs) other than acetylsalicylic acid is prohibited.
    * Selective serotonin reuptake inhibitors or selective serotonin norepinephrine reuptake inhibitors, if a subject is not compliant with the medication and/or has not been receiving a stable dose for at least 3 months prior to Screening.
    * Tricyclic antidepressants, if a subject is not compliant with the medication and/or has not been receiving a stable dose for at least 3 months prior to Screening.
    * Any angiotensin vaccine, including prior exposure to ATV.
20. Have participated in a clinical study involving another investigational drug or device within 4 weeks of Screening.
21. Any concomitant condition that, in the opinion of the investigator, may adversely affect the safety and/or efficacy of the study drug or severely limit the subject's ability to complete the study (eg, disabling or terminal illness, mental disorders).
22. Any major contraindication to stopping antihypertension medications for a period of up to 14 weeks.
23. Previous exposure to CoVaccine HT adjuvant, or other keyhole limpet haemocyanin-containing vaccines.
24. Previous serious reaction to a vaccine, such as angioedema or anaphylaxis.
25. Known history of drug and/or alcohol abuse and those known to be hepatitis positive.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wajdi H Turkie, MD, Principal Investigator — The Acumen Pharmaceuticals Services Ltd
Locations (12):
- United Kingdom (12):
  - Fowey River Practice, Fowey, Cornwall
  - Alverton Practice, Penzance, Cornwall
  - Brannel Surgery, Saint Stephen, Cornwall
  - Saltash Health Centre, Saltash, Cornwall
  - Cape Cornwall Surgery, St Just, Cornwall
  - Avondale Surgery, Chesterfield, Derbyshire
  - Knowle House Surgery, Plymouth, Devon
  - Layton Medical Centre, Blackpool, Lancashire
  - Sherbourne Medical Centre, Royal Leamington Spa, Warwickshire
  - Abbey Meads Medical Practice, Swindon, Wiltshire
  - Grey Gable Surgery, Inkberrow, Worcestershire
  - The Acumen Pharmaceutical Services Ltd, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Investigators provide information to participants

RESULTS

PARTICIPANT FLOW:
Groups:
- Angiotensin Therapeutic Vaccine With CoVaccine HT™ Adjuvant: Angiotensin Therapeutic Vaccine with CoVaccine HT™ adjuvant (an ingredient that may improve the immune response of the vaccine)
  Angiotensin Therapeutic Vaccine plus CoVaccine HT™ adjuvant: Given as three separate intramuscular injections into the arm, 21 days apart
- CoVaccine HT™ Adjuvant Alone (Control): CoVaccine HT™ adjuvant alone
  CoVaccine HT™ adjuvant: Given as three separate intramuscular injections into the arm, 21 days apart
Period: Overall Study
Arm/Group | Angiotensin Therapeutic Vaccine With CoVaccine HT™ Adjuvant | CoVaccine HT™ Adjuvant Alone (Control)
Started | 10 | 10
Completed | 6 | 7
Not Completed | 4 | 3
Not completed — Adverse Event | 4 | 3

BASELINE CHARACTERISTICS:
Population: All analyzed subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Angiotensin Therapeutic Vaccine With CoVaccine HT™ Adjuvant | CoVaccine HT™ Adjuvant Alone (Control) | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (6.94) | 53.7 (6.63) | 52.8 (6.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Mean Daytime Diastolic Blood Pressure (DBP) Measured by Ambulatory Blood Pressure Monitoring (ABPM)
Time Frame: baseline to 8 weeks
Population: study prematurely terminated
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Angiotensin Therapeutic Vaccine + CoVaccine HT™ Adjuvant: Angiotensin Therapeutic Vaccine + CoVaccine HT™ adjuvant (an ingredient that may improve the immune response of the vaccine)
  Angiotensin Therapeutic Vaccine + CoVaccine HT™ adjuvant: Given as three separate intramuscular injections into the arm, 21 days apart
Arm/Group | Angiotensin Therapeutic Vaccine + CoVaccine HT™ Adjuvant | CoVaccine HT™ Adjuvant Alone (Control)
Number analyzed (Participants) | 6 | 7
mmHg | -7.18 (3.451) | -3.68 (3.049)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Angiotensin Therapeutic Vaccine With CoVaccine HT™ Adjuvant | CoVaccine HT™ Adjuvant Alone (Control)
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angiotensin Therapeutic Vaccine With CoVaccine HT™ Adjuvant (N=10) | CoVaccine HT™ Adjuvant Alone (Control) (N=10)
cellulitis (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Angiotensin Therapeutic Vaccine With CoVaccine HT™ Adjuvant (N=10) | CoVaccine HT™ Adjuvant Alone (Control) (N=10)
injection site pain (General disorders) | 9 (9) | 8 (8)
chills (General disorders) | 4 (4) | 3 (3)
pain (General disorders) | 2 (2) | 0 (0)
headache (Nervous system disorders) | 9 (9) | 6 (6)
hyperesthesia (Nervous system disorders) | 1 (1) | 0 (0)
tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
cellulitis (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study prematurely terminated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No